CLINICAL TRIAL: NCT06313177
Title: Syndesmotic Screw in Neutral Position Versus Maximum Ankle Dorsiflexion in Ankle Fractures; Comparative Study.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Asaad Mahmoud, Resident-orthopedic department-sohag hospital university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Soh-Med-24-03-03MS
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Syndesmotic Injuries
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): group(A) cases with ankle in neutral position during syndesmosis fixation
  Interventions: Procedure: syndesmosis fixation with screws
- group B (Active Comparator): group(B) cases with ankle in dorsiflexion position during syndesmosis fixation
  Interventions: Procedure: syndesmosis fixation with screws

INTERVENTIONS:
Procedure: syndesmosis fixation with screws — syndesmosis fixation with Syndesmotic screw in neutral position versus maximum ankle dorsiflexion in ankle fracture

SUMMARY:
Ankle fracture is one of the most common orthopedic injuries. Approximately, 20% of surgically treated ankle fractures are associated with syndesmotic instability.According to the mechanism of the injury the syndesmotic disruption should be considered in Danis-Weber C-type fractures. However, such injuries were also frequently seen in Danis-Weber B-type fractures. Failure to detect and repair syndesmotic injuries early may result in poor clinical outcomes and complications affecting ankle function, such as long-term residual pain, post traumatic arthritis, and ankle impingement syndromes. Therefore, aggressive treatment is important when facing syndesmotic instability .

The distal tibiofibular syndesmosis is important for stability of the ankle mortise and thus for weight transmission and walking. Syndesmotic injuries are most commonly associated with fibular fractures, but they can also occur in isolation or with damage to the lateral ankle ligament after traumatic supination. The need for syndesmotic fixation of the distal tibiofibular joint has been controversia. fracture does not correlate reliably with the extent of the interosseous membrane tears identified on MRI of ankle fractures, and thus estimation of the integrity of the interosseous membrane and subsequent need for trans-syndesmotic fixation cannot be based solely on the level of the fibular fracture. An intraoperative syndesmotic stress test can establish the presence or absence of syndesmotic instability, evaluating the integrity of the syndesmosis by grasping the stabilised fibula with a hook or clamp and pulling it laterally. If more than 3 or 4 mm of lateral displacement occurs, syndesmotic fixation is necessary.

Most authors recommend surgical placement of a trans-fixation screw after anatomical reduction of the syndesmosis if a disruption is diagnosed to avoid complications.The main aims of treatment for dislocation of the distal tibiofibular syndesmosis are to restore the original anatomy and normal function and to recreate the stability of the ankle joint. The syndesmosis is traditionally fixed with a metallic screw, which is a method that has been used for decades and demonstrates good to excellent outcomes.

Some surgeons prefer Fixation of syndesmosis with screw in maximum ankle dorsiflexion and others prefer fixation in neutral position of ankle.in this study we are going to compare between these two

ELIGIBILITY:
Inclusion Criteria:

* patients with fracture Ankle type C and type B associated with syndesmotic injury

Exclusion Criteria:

* pathologic fractures
* Maisonneuve fractures
* medical illness or mental disorders affecting the follow-up examination
* loss to follow-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-10 (Estimated); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
pain with AOFAS score | 1 year
  The AOFAS ankle-hindfoot score is a clinical rating system associated patients-reported outcomes with clinician-measured outcomes to make a 100-point scale that comprises nine questions in approximately three categories: pain (one question; 40 points), function (seven questions; 50 points) and alignment (one question; 10 points). Through this questionnaire, the condition of the ankle could be described in a more comprehensive and simple way

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Zuuren WJ, Schepers T, Beumer A, Sierevelt I, van Noort A, van den Bekerom MPJ. Acute syndesmotic instability in ankle fractures: A review. Foot Ankle Surg. 2017 Sep;23(3):135-141. doi: 10.1016/j.fas.2016.04.001. Epub 2016 Apr 25. PMID 28865579
- [Background] Cornu O, Manon J, Tribak K, Putineanu D. Traumatic injuries of the distal tibiofibular syndesmosis. Orthop Traumatol Surg Res. 2021 Feb;107(1S):102778. doi: 10.1016/j.otsr.2020.102778. Epub 2020 Dec 14. PMID 33333279
- [Background] Corte-Real N, Caetano J. Ankle and syndesmosis instability: consensus and controversies. EFORT Open Rev. 2021 Jun 28;6(6):420-431. doi: 10.1302/2058-5241.6.210017. eCollection 2021 Jun. PMID 34267932
- [Background] Kitaoka HB, Alexander IJ, Adelaar RS, Nunley JA, Myerson MS, Sanders M. Clinical rating systems for the ankle-hindfoot, midfoot, hallux, and lesser toes. Foot Ankle Int. 1994 Jul;15(7):349-53. doi: 10.1177/107110079401500701. PMID 7951968